CLINICAL TRIAL: NCT06476639
Title: A Phase III Randomised Clinical Trial of Ultrasound Groin Monitoring Versus Groin Lymph Node Dissection to De-Escalate the Extent of Surgery in Vulvar Cancer
Acronym: ANVU
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANVU
Record Dates: First submitted 2024-06-17; First posted 2024-06-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Vulvar Cancer Stage I; Vulvar Cancer Stage II; Lymph Node Metastasis; Groin Node; Ultrasound Therapy; Complications
Keywords: Vulvar Cancer; Ultrasound Therapy
MeSH Terms: conditions — Vulvar Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Intervention Model Description: A phase III, open label, multicentre, three-group, randomised clinical trial.
  640 eligible females aged 18 or older with clinically stage 1b or 2 vulvar cancer will receive a bilateral groin node ultrasound up to 30 days prior to planned surgery:
  Participants with normal/negative baseline groin ultrasounds will be randomly assigned to two groups (3:1 randomisation). The Intervention Group will receive serial bilateral groin node ultrasounds and clinical examinations for 18 months (groin lymph nodes are not removed). The Standard Group will undergo upfront full groin lymph node dissection (LND) or sentinel node biopsy (SNB) based on clinician choice (according to local clinical practice management guidelines).
  Participants with abnormal baseline groin ultrasound (third group) will receive an upfront full groin LND or SNB, consistent with the current standard treatment, according to local clinical practice management guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participants with normal/negative baseline groin ultrasounds - Intervention Group (Experimental): Surgical removal of primary tumour and serial high-resolution bilateral groin ultrasound monitoring every 2 months for 12 months, and at month 15 and month 18, with clinical examination at 8 weeks, 4 months, 8 months, 12 months, 15 months, and 18 months (n=360).
  Interventions: Diagnostic Test: High-resolution bilateral groin ultrasound monitoring
- Participants with normal/negative baseline groin ultrasounds - Standard Group (No Intervention): Surgical removal of primary tumour and upfront full groin lymph node dissection (LND) or sentinel node biopsy (SNB) based on clinician choice (according to local clinical practice management guidelines) (n=120).
- Participants with suspicious/indeterminate baseline groin ultrasound - Standard Treatment (No Intervention): Participants with suspicious/indeterminate baseline groin ultrasound (third group) will receive an upfront full groin LND or SNB, consistent with the current standard treatment, according to local clinical practice management guidelines (n=160).

INTERVENTIONS:
Diagnostic Test: High-resolution bilateral groin ultrasound monitoring — Participants in the Interventional Group will undergo surgical excision of the primary tumour, either via radical local excision or radical vulvectomy. Post-vulvar surgery, participants will receive a groin node ultrasound every 2 months for 12 months, and at month 15 and month 18, and a clinical examination at 8 weeks, 4 months, 8 months, 12 months, 15 months, and 18 months. Senior imaging specialists review bilateral ultrasound scans for positive lymph nodes or suspicious findings, promptly sending reports to the primary care physician and trial manager within 5 business days. If positive nodes are detected, participants will consult their primary care physician for options. Depending on clinical judgment, they may be referred for LND or continue with serial ultrasounds and clinical exams based on preference and clinician guidance.
  Arms: Participants with normal/negative baseline groin ultrasounds - Intervention Group

SUMMARY:
This study is a phase III, open label, multicentre, three-group, randomised clinical trial. The primary aim of this study is to determine whether intensive groin ultrasound monitoring (1) is effective and safe to replace invasive groin lymph node dissection (LND) to manage vulvar cancer, (2) decreases the morbidity associated with vulvar cancer surgery, and (3) is cost effective.

DETAILED DESCRIPTION:
Treatment of vulvar cancer causes significant morbidity. Despite being a rare cancer, at least 2500 survivors of vulvar cancer live in Australia. Most survivors live with the detrimental, life-long impacts resulting from their cancer treatment because there are currently no alternatives to mitigate these impacts. The personal and societal burden this entails is significant. To control such cancer-associated burden is a national priority.

Clinical palpation of the groin region and computed tomography (CT) scans do not reliably detect groin node involvement. Hence, current clinical guidelines recommend all women diagnosed at apparent Stage I or II have a surgical groin LND. This can be performed as a full IFL (full LND) to remove all groin nodes, or as a sentinel node biopsy (SNB) to remove selected (one or two) nodes. SNB is less invasive, however, is appropriate only for vulvar cancers <4cm in diameter and unifocal tumours (~50% of all Stage I and II vulvar cancers). SNB is also associated with a false negative rate (10%) that increases the risk of undetected nodes.

In 25% of cases (~80 Australian women per year), groin LND will reveal positive nodes (i.e., metastases), which triggers a referral for radiation treatment. If positive groin nodes are missed, and over time become enlarged, clinically palpable and attached to the overlying skin, >90% of women will die within 12 months, despite subsequent treatment. Conversely, if groin node involvement is detected early (e.g., by ultrasound) while still small, survival outcomes are excellent. Ultrasound technology is potentially as accurate as LND due to recent advances in resolution and technologies such as 2D/3D volumetric assessments and tissue flow. Furthermore, ultrasound is superior to medical resonance imaging (MRI), and to standard CT and positron emission tomography (PET) scans in capturing groin node involvement because it has a higher resolution, avoids harmful radiation and the technology is readily accessible outside of high-volume metropolitan areas.

The investigators propose to reduce surgical morbidity by replacing upfront groin LND for vulvar cancer patients with serial high-resolution ultrasound to detect groin metastases. Groin LND will only be necessary for the few women with ultrasound-detected metastases when they are still small. The ANVU trial will determine the value of serial groin ultrasound examinations in stage 1b and 2 vulvar cancer patients and whether it is feasible and safe to de-escalate the extent of vulvar cancer surgery to achieve improved outcomes for affected patients.

Women with this rare cancer bear an unacceptably high (and potentially avoidable) treatment-related burden. This clinical trial is the first step to address this problem in a novel yet pragmatic way. The potential overall outcome of ANVU could be a novel, less invasive alternative to vulvar cancer LND hypothesised to be associated with significantly less morbidity, without compromising survival.

ELIGIBILITY:
Inclusion Criteria:

* Females, over 18 years, with histologically confirmed SCC or adenocarcinoma of the vulva
* Clinically stage 1b or 2 on medical imaging (CT or MRI scan of pelvis, abdomen, and chest), without evidence of regional or distant metastatic disease
* Willing and able to undergo IFL/SNB according to local clinical practice management guidelines
* Willing and able to comply with all study requirements, timing and/or nature of required assessments.
* Signed written informed consent
* Negative (serum or urine) pregnancy (BHCG) test ≤ 30 days of surgery ONLY in pre-menopausal women and women < 2 years after the onset of menopause.

Exclusion Criteria:

* Women with non-invasive vulvar conditions (e.g. non-invasive non-mammary Paget's disease)
* Clinical or medical imaging evidence of regional and/or distant metastatic disease
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
* Other prior malignancies <5 years before inclusion, except for successfully treated keratinocyte skin cancers, or ductal carcinoma in situ
* Estimated life expectancy of ≤6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 640 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Death secondary to the development of groin node metastasis (GND, Groin Node-related Death) at 30 months. | 30 months
  Determine the risk of death secondary to the development of groin node metastasis (GND, Groin Node-related Death) in patients with vulvar cancer randomised to serial high-resolution groin USM compared to standard upfront surgical groin LND at 30 months.

SECONDARY OUTCOMES:
Compare return to usual daily activities at 18 months between the groups | 18 months
  Return to usual daily activities at 18 months measured using the PROMIS Ability to Participate in Social Roles and Activities Short Form 8a
HRQL and PROMS as measured by the EQ-5D and FACT-V at baseline, 8 weeks, 6 months, 12 months, 18 months, 24 months, and 30 months. | 30 months
  Compare Patient Reported Outcomes (PROMs) and Health Related Quality of Life (HRQL) between the groups.
Morbidity at 12 months after surgery. | 12 months
  Compare pain and adverse events (AEs) (morbidity) between the groups.
Incidence of lower limb lymphoedema up to 30 months after surgery. | 30 months
  Compare the incidence of lower limb lymphoedema at 30 months post-surgery between the groups.
Cost and cost-effectiveness at 12 months post-surgery. | 12 months
  Compare cost and cost-effectiveness between the groups.
Fear of recurrence at baseline, 8 weeks, 6 months, 12 months, 18 months, 24 months, and 30 months. | 30 months
  Compare fear of recurrence between the groups.
Clinical accuracy of high-resolution ultrasound to predict groin lymph node involvement. | 18 months
  Determine the diagnostic accuracy of standardised, high-resolution groin ultrasound to identify groin node metastasis.
Disease-free survival (DFS) and overall survival (OS) at 30 months. | 30 months
  Compare disease free and overall survival between the groups.
Determine compliance with serial ultrasound scans. | 18 months
  Compliance with serial ultrasound scans.
Utility of biomarkers to reliably reflect the presence or absence of positive groin lymph nodes, and explore novel biomarkers for vulvar cancer. | Up to 15 years
  Assess the role of blood and tissue molecular biomarkers to accurately determine the burden of disease (positive lymph nodes) in vulvar cancer, assist with risk stratification and aid disease surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, MD, Study Chair — Director, Queensland Centre for Gynaecological Cancer Research
Locations (9):
- Australia (9):
  - John Hunter Hospital, Newcastle, New South Wales
  - The Royal Darwin Hospital, Darwin, Northern Territory
  - The Wesley Hospital, Auchenflower, Queensland
  - St Andrew's War Memorial Hospital, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Buderim Private Hospital, Buderim, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Mercy Hospital for Women, Heidelberg, Victoria
  - Royal Women's Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No